CLINICAL TRIAL: NCT04837846
Title: Multicenter Study Into Individualized Scanning for Coronary Artery Disease
Acronym: MINDS-CAD
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 00093255
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective CCTA Arm
  Interventions: Other: Differing Tube Voltage Administration

INTERVENTIONS:
Other: Differing Tube Voltage Administration — Subjects will undergo CCTA utilizing a scan and contrast media injection protocol that will be tailored to individual body habitus.

SUMMARY:
To evaluate intravascular attenuation of the coronary arteries and image quality in an individualized scan and CM injection protocol whereas both scan and injection parameters are tailored to the individual patient in a North American, European and Asian patient population.

To evaluate the radiation dose and contrast media dose of this individualized approach for CCTA in an American, European and Chinese patient population.

To evaluate the injection parameters required for an average American, European and Chinese patient population.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study: (All answers must be "YES" for subject to be eligible.)

  1. Referred for a clinically indicated CCTA scan.
  2. Patient aged older than 18.
  3. Subject must provide written informed consent prior to any study-related procedures being performed.
  4. Subject must be willing to comply with all clinical study procedures.
  5. Atypical or typical complaints of angina.
  6. No previous cardiovascular history.
  7. Possibility of 'flash' mode scan; patient heart rate below 70 beats per minute and regular rhythm.

Exclusion Criteria:

* The presence of the following excludes subjects from the study: (All answers must be "NO" for subject to be eligible.)

  1. Contraindications for CT coronary angiography, including:

     1. Inability to perform a breath hold for at least the expected scan time
     2. Unstable angina
     3. Hemodynamic instability
     4. Known history of CAD
     5. Pregnancy
     6. Renal insufficiency (defined as Creatinine <1.5 mg/dL or GFR<30 mL/min)
     7. Iodine allergy
  2. Insufficient cannula venous access (preferred 18G, minimal 20G cannula)
  3. Subject has an acute psychiatric disorder.
  4. Subject is unwilling to comply with the requirements of the protocol.
  5. Subject has previously entered this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with complaints of angina, referred for a clinically indicated CCTA scan
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of Intravascular Attenuation | At time of CCTA scan
  To measure the amount of Hounsfield units in different anatomical structures produced by an amount of contrast media. Using Hounsfield units coupled with image quality to determine if a scan of diagnostic value has been attained.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph U. Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes